CLINICAL TRIAL: NCT02124187
Title: Smoking Cessation And Reduction in Depression
Acronym: scarid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universita degli Studi di Catania (Other)
Collaborators: Lega Italiana Anti Fumo (Other)
Responsible Party: Principal Investigator, Riccardo Polosa, Full Professor of internal medicine, Universita degli Studi di Catania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCARID
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Tobacco Smoking in Depressed Patients
MeSH Terms: interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- eCig 24 mg nicotine (Experimental): eCig 24 mg nicotine for 12 weeks
  Interventions: Device: Ecig 24 mg nicotine
- Ecig 0 mg nicotine (Sham Comparator): eCig 0 mg nicotine for 12 weeks
  Interventions: Device: Ecig 0 mg nicotine
- Nicotine free inhalator (Placebo Comparator): nicotine free inhalator for 12 weeks
  Interventions: Device: Nicotine free inhalator

INTERVENTIONS:
Device: Ecig 24 mg nicotine — eCig 24 mg nicotine for 12 weeks
  Arms: eCig 24 mg nicotine
Device: Ecig 0 mg nicotine — eCig 0 mg nicotine for 12 weeks
  Arms: Ecig 0 mg nicotine
Device: Nicotine free inhalator — eCig 24 mg nicotine for 12 weeks
  Arms: Nicotine free inhalator

SUMMARY:
It is well established in studies across several countries that tobacco smoking is more prevalent among depressed patients than the general population. Electronic cigarettes are becoming increasingly popular with smokers worldwide. To date there are no large randomized trials of electronic cigarettes in depressed smokers. A well-designed trial is needed to compare efficacy and safety of these products in this special population.

We have designed a randomized controlled trial investigating the efficacy and safety of electronic cigarette. The trial will take the form of a prospective 12-month randomized clinical study to evaluate smoking reduction, smoking abstinence and adverse events in depressed smokers not intending to quit. We will also monitor quality of life, neurocognitive functioning and measure participants' perception and satisfaction of the product.

Outcome measures: A ≥50% reduction in the number of cigarettes/day from baseline, will be calculated at each study visit ("reducers"). Abstinence from smoking will be calculated at each study visit ("quitters"). Smokers who leave the study protocol before its completion and will carry out the Early Termination Visit or who will not satisfy the criteria of "reducers" and "quitters" will be defined "non responders".

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Major Depressive Disorder (MDD) (according to DSM 5 criteria) from throughout Sicily (Italy), who smoke tobacco cigarettes.
2. smoke ≥10 factory made cig/day, for at least the past five years
3. age 18-65 years
4. in good general health (in absence of cancer, acute myocardial infarction, unstable angina, severe cardiac arrhythmia, recent cerebrovascular incident, or severe atherosclerosis )
5. not currently attempting to quit smoking or wishing to do so in the next 30 days (a specific test will be included to check their unwillingness to quit) 6 months
6. committed to follow the trial procedures.

Exclusion Criteria:

1. use of smokeless tobacco or nicotine replacement therapy or other smoking cessation therapies
2. pregnancy or breastfeeding
3. current or recent (less than 1 yr) past history of alcohol and/or drug abuse
4. active suicidal intention
5. other significant co-morbidities according to the Investigator's clinical assessment (e.g. cancer, acute myocardial infarction, unstable angina, severe cardiac arrhythmia, recent cerebrovascular incident, or severe atherosclerosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Smoking Cessation | 52 weeks
  Abstinence from smoking, defined as complete self-reported abstinence from tobacco smoking - not even a puff (together with an eCO concentration of ≤7 ppm), will be calculated at each study visit ("quitters").

SECONDARY OUTCOMES:
Smoking reduction | 52 weeks
  A ≥50% reduction in the number of cig/day from baseline, defined as self-reported reduction in the number of cig/day (≥50%) compared to baseline (together with an eCO levels reduction, to objectively document a reduction from baseline), will be calculated at each study visit ("reducers").

OTHER OUTCOMES:
Neuro cognitive functioning and product preferencies | 52 weeks
  Quality of life, Neurocognitive Functioning and Psychopathological status will be reassessed by Quality of Life Scale (QLS), Repeatable Battery for the assessment of Neuropsychological Study (RBANS) and Hamilton Depression Rating Scale (HDRS), respectively.
  Participants' perception and liking of the product will be assessed by asking to rate their level of satisfaction with the products compared to their own cigarettes using a visual analogue scale (VAS) from 0 to 10 points (0 = being 'completely unsatisfied', 10 being = 'fully satisfied'); using the same scale, they will also rate how much they miss their own brand (0 = being 'did not miss it at all', 10 being = 'missed too much') and whether they would recommend it to a friend/relative (0 = being 'not recommended at all', 10 being = 'absolutely recommended').

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Policlinico - Vittorio Emanuele di Catania, Catania, Sicily, Italy

REFERENCES:
- [Background] Caponnetto P, Polosa R, Auditore R, Minutolo G, Signorelli M, Maglia M, Alamo A, Palermo F, Aguglia E. Smoking cessation and reduction in schizophrenia (SCARIS) with e-cigarette: study protocol for a randomized control trial. Trials. 2014 Mar 22;15:88. doi: 10.1186/1745-6215-15-88. PMID 24655473